CLINICAL TRIAL: NCT04732013
Title: Nonselection Pilot Study to Assess the Clinical Efficacy of Noninvasive Preimplantation Genetic Testing for Aneuploidy
Brief Title: Noninvasive Chromosomal Screening for Embryo Selection Trial
Acronym: NICEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Olive Fertility Centre (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry); Sequence46 (Unknown)
Responsible Party: Principal Investigator, Gary Nakhuda, Co-Director, Olive Fertility Centre
Other Study IDs: NI-PGTA
Record Dates: First submitted 2020-11-27; First posted 2021-02-01 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Infertility; Aneuploidy
Keywords: IVF; PGT-A; Aneuploidy
MeSH Terms: conditions — Infertility; Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Spent culture media from cultured blastocysts which is typically discarded will be collected to isolate free DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Single observational cohort of patients who meet study criteria
  Interventions: Other: No clinical intervention is planned; study is observational

INTERVENTIONS:
Other: No clinical intervention is planned; study is observational — No intervention

SUMMARY:
To determine the diagnostic accuracy of non-invasive preimplantation genetic testing for aneuploidy (NI-PGT-A) for embryo selection.

DETAILED DESCRIPTION:
Hypothesis:

Analysis of cell free DNA (cfDNA) released from developing embryos into spent culture media (SCM) can serve as a non-invasive method for performing preimplantation genetic testing for aneuploidy (PGT-A). A non-selection study that compares clinical outcomes to the NI-PGT-A results of the transferred embryos in a blinded fashion will characterize the diagnostic accuracy by determination of positive and negative predictive values

Justification:

During the in vitro fertilization (IVF) process, the selection of a healthy embryo is limited by the inability of the microscopic appearance to reveal the chromosomal complement. Thus, in order to reliably select chromosomally normal embryos, preimplantation genetic testing for aneuploidy (PGT-A) is performed. PGT-A requires biopsy of the embryo, amplification of the DNA, then next generation sequencing (NGS) to determine chromosome copy number.

While the clinical utility of PGT-A has been demonstrated, the process has limitations, the most significant of which is the requirement for embryo biopsy. Typically, 5-10 cells are removed from the TE after the zona pellucida has been breached. While the procedure can be safely and effectively performed by trained embryologists, the obvious concern for damage to the embryo is relevant. Even if implantation successfully occurs, concern has been raised that biopsy of the embryo at this stage can lead to complications such as miscarriage, or issues with placental function later in pregnancy. Furthermore, because the TE is destined to differentiate to placenta rather than the fetus itself, there is controversy regarding if the chromosomal analysis of these cells is always representative of the chromosomal complement of the fetus. For these reasons, and because TE biopsy is laborious and expensive, PGT-A has still not supplanted morphological evaluation as the clinical standard for embryo selection.

An accurate noninvasive method for aneuploidy screening of embryos before implantation would be ideal. To this end, development of noninvasive PGT-A (NI-PGT-A) methods is an area of active investigation. The approach leverages the ability to isolate cell-free DNA (cfDNA) that is secreted from the blastocyst into the spent culture media (SCM). SCM is routinely discarded after the embryo has been removed from culture, however, minute amounts of DNA from the embryo can be isolated, amplified, then sequenced for chromosomal copy number analysis. The obvious advantage is that this process can occur without posing any harm to the embryo. An additional putative benefit of this noninvasive approach is that the DNA is secreted from both the TE and the inner cell mass (ICM), theoretically serving as a more accurate representation of the fetal karyotype than the DNA isolated from just the TE biopsy alone.

Technical limitations of deploying NI-PGT-A are related to the limited quantity of DNA available in the SCM. Unlike other modes of genetic testing where ample amounts of genetic material is readily extracted from blood, amniotic fluid, or tissue biopsy, cell-free DNA secretion from blastocysts is exceptionally minute in quantity. However, laboratory protocols are developing rapidly, evidenced by numerous publications which have already demonstrated a high level of consistency when chromosomal copy number is analyzed by NI-PGT-A and traditional PGT-A in parallel.

While these studies have illustrated proof of concept and preclinical validation, the true diagnostic accuracy can only be assessed by evaluating the predictive value of negative (euploid) and positive (aneuploid) results. Specifically, embryos found to be euploid should have a greater ability for sustained implantation that proceeds to live birth, while aneuploid embryos should have a dramatically lower rate of sustained implantation, or will be predictive of clinical aneuploidy. Without rigorous clinical validation, using these results for embryo selection could lead to misdiagnosis, causing selection of unhealthy embryos, or selection against embryos that could have been potentially viable.

To determine if NI-PGT-A is clinically robust, we propose a non-selection, pilot, study, whereby embryo selection is performed by routine clinical methods (ie, morphological selection). However, after the clinical outcome has manifested, the SCM will be analyzed by a commercially available NI-PGT-A protocols in a blinded fashion. By correlating clinical outcomes to NI-PGT-A results, positive and negative predictive values can be calculated without bias. Because no intervention will be performed that deviates from the clinical routine, no additional risk will be posed to the embryo or parent.

This study will serve as a pilot for a possible future trials. If reasonable predictive value of NI-PGT-A is demonstrated, a prospective, selection study could be justified to investigate the utility of NI-PGT-A in a clinical setting.

Research Design:

Patients will undergo IVF-ICSI per clinical indication, with plans to freeze all embryos for deferred embryo transfer. Embryo culture will follow routine protocols and embryo selection for transfer will be performed using standard morphological criteria. SCM from all blastocysts that appear viable will be collected and shipped to a reference lab (Sequence 46). Specimens will be completely de-identified of patient information and labelled with an accession number. NI-PGT-A analysis will be performed using a commercial kit according to manufacturer's recommendations, with technicians blinded to clinical outcomes. When patients return for the embryo transfer cycle, routine clinical protocol will be followed for endometrial preparation. A single embryo will be selected according to routine morphological grading criteria, and embryo transfer will be performed with standard techniques. Initial pregnancy outcome will be documented with serum hCG testing. If hCG testing is positive, early pregnancy will be confirmed with ultrasound assessment per clinical routine. After all patients have completed treatment and clinical outcomes manifested (failed implantation, miscarriage, or ongoing pregnancy (defined as viability beyond 13 weeks), NI-PGT-A results will be released to the clinical team and correlated to clinical outcomes for calculation of predictive values. All on-going pregnancies will be offered routine prenatal screening for fetal aneuploidies.

Additional details regarding laboratory protocols are as follows:

Blastocyst culture Embryo culture will follow routine protocols. On day 3 post-fertilization, embryos will be repeatedly pipetted through a series of culture media droplets in order to lower potential for maternal cell contamination. Embryos will then be individually cultured in 35µL droplets of embryo culture medium to the blastocyst stage. On day 5 or day 6, blastocyst development and quality will be evaluated using standard morphological criteria.

Sample collection and blastocyst vitrification Blastocyst culture medium (20µL) from selected embryos will be collected and transferred to PCR tubes and stored at -20°C until whole genome amplification (WGA). Blastocysts will be frozen via routine vitrification protocol and stored in liquid nitrogen per routine clinical protocol. Specimens will be completely de-identified of patient information and labelled with an accession number prior to shipping to reference lab (Sequence46).

Whole genome amplification and DNA sequencing NI-PGT-A analysis will be performed upon receipt, using a commercial kit according to manufacturer's recommendations, with technicians blinded to clinical outcomes. DNA will be amplified by whole genome amplification (WGA) and barcoded to prepare libraries. The libraries are then loaded onto an Ion Chef instrument for template preparation by automated clonal amplification and then loaded onto a chip for DNA sequencing on an Ion Genestudio S5 Prime system, with approximately 150,000-200,000 sequencing reads per sample. Data is analyzed using the Ion Reporter software (v5.10 or later). Ploidy will be measured using baseline, Ion ReproSeq Low-Coverage Whole-Genome (99M) Baseline. Standard quality control measures will be evaluated. Results will be released to the clinical team 6 weeks post-embryo transfer and correlated to clinical outcomes for calculation of predictive values.

Patient population:

Inclusion Criteria:

Patient undergoing IVF-ICSI 21 - 35 years old at the time of enrollment Elective freeze-all cycle Planning for single embryo transfer

Exclusion Criteria:

Undergoing PGT-A, PGT-SR, PGT-M History of recurrent pregnancy loss History of recurrent implantation failure Planning on transfer of more than 1 embryo

The justification for the age category is to control for age-related factors other than aneuploidy that may influence implantation, so variables that could compound predictive value calculations are minimized. Limiting participation to patients under 35 also optimizes embryo selection such that morphologically normal embryos are most likely healthy. Furthermore, patients in this age category have the lowest risk for clinical aneuploidies such as Down syndrome.

Data management and storage:

Research samples will be identified by a unique accession number, but no patient identifying information. The samples will be processed by Sequence46 with results associated with the accession number. The data will be uploaded via a secure cloud service, which will be accessed by the primary investigator to merge with the electronic case report form (eCRF) that will be stored locally at the Olive Fertility Centre on an encrypted hard drive that will be backed-up on a secondary local drive. The eCRF will contain the patients' unique medical record number and age, but will not document name, birthdate, or any other identifying information. Results of the NI-PGT-A analysis and clinical outcome will also be stored in the eCRF.

Research data will be retained for 5 years after the date of publication.

Statistical analysis:

Diagnostic accuracy will be interpreted in the context of positive and negative predictive values.

A positive result is a finding consistent with aneuploidy or mosaicism. A negative result is a finding consistent with euploidy.

PPV = (Failed implantation + miscarriage + clinical aneuploidy)/ All Positive Results NPV = Ongoing pregnancy / All Negative Results

Sample size calculation:

One hundred-twenty (120) patients should suffice for this pilot study. Previous research has established that in patients aged 35 or younger, the ratio of euploid:aneuploid embryos is approximately 60:40. Of euploid embryos, approximately 70% will implant, of which, 85% should continue to viability. Of aneuploid embryos, approximately 25% will implant, of which >99% will miscarry; the risk of a clinical aneuploidy is less than 0.5% in women 35 and under.

Given these probabilities, of the 120 patients to be enrolled, 72 euploid embryos are expected of which 50 should implant and 43 will continue as ongoing, viable pregnancies. Of the 48 that are expected to be aneuploid, 12 will implant, of which all should miscarry (the chance for a clinical aneuploidy in this population is less than 0.5%).

Recruitment:

Patients who are pursuing IVF-ICSI at the Olive Fertility Centre and meet inclusion/exclusion criteria will be recruited directly by the co-investigators. Flyers will be posted within the clinic.

ELIGIBILITY:
Inclusion Criteria:

Patient undergoing IVF-ICSI at the Olive Fertility Centre

* 21 - 35 years old at the time of enrolment
* Elective freeze-all cycle
* Planning for single embryo transfer

Exclusion Criteria:

* Undergoing PGT-A, PGT-SR, PGT-M
* History of recurrent pregnancy loss
* History of recurrent implantation failure
* Planning on transfer of more than 1 embryo

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing IVF-ICSI at the Olive Fertility Centre that fit the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-09-04 (Estimated); Study Completion 2022-12-04 (Estimated)

PRIMARY OUTCOMES:
Predictive value of NI-PGT-A results with implantation rate. | 1 year
  Positive and negative predictive value of NI-PGT-A results to embryo implantation rate determined by quantitative hCG levels and ultrasound findings.
Predictive value of NI-PGT-A results with on-going pregnancy rate. | 1 year
  Positive and negative predictive values of NI-PGT-A results with ongoing pregnancy rates as determined by viability through the 1st trimester.
Predictive value of NI-PGT-A results with miscarriage rate. | 1 year
  Positive and negative predictive values of NI-PGT-A results with miscarriage rates documented in the 1st trimester.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Nakhuda, MD, Principal Investigator — Olive Fertility Centre
Locations (1):
- Olive Fertility Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nakhuda G, Rodriguez S, Tormasi S, Welch C. A pilot study to investigate the clinically predictive values of copy number variations detected by next-generation sequencing of cell-free deoxyribonucleic acid in spent culture media. Fertil Steril. 2024 Jul;122(1):42-51. doi: 10.1016/j.fertnstert.2024.02.030. Epub 2024 Feb 19. PMID 38382698